CLINICAL TRIAL: NCT04915976
Title: Gender-specific Temporal Trends in Survival in Patients With Severe Aortic Stenosis Undergoing Transfemoral Transcatheter Aortic Valve Implantation.
Brief Title: TAVI and Gender Outcomes Aortic Stenosis Undergoing Transfemoral Transcatheter Aortic Valve Implantation.
Status: Suspended | Type: Observational
Why Stopped: Dataset not obtained
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Ghada Mikhail, Consultant Cardiologist, Imperial College Healthcare NHS Trust
Other Study IDs: 283163
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Aortic Stenosis; Gender; Surgery
Keywords: aortic stenosis, TAVR, TAVI, Transcatheter aortic valve implantation, Gender differences
MeSH Terms: conditions — Aortic Valve Stenosis; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe aortic stenosis (AS) is the commonest form of valvular abnormality in the developed world and transcatheter aortic valve implantation (TAVI) is now widely practiced as in many cases is the preferred treatment option over conventional aortic surgery. Several studies have shown that females have an apparent better outcome with TAVI than males.

There are a number of possible reasons as to the apparent favourable benefit of TAVI in women including: having both lower rates of moderate / severe aortic regurgitation and peri-procedural mortality, lower rates of bleeding and renal failure, better patient prosthesis match and recovery of left ventricular function with more favourable left ventricular remodelling.

We aim to explore the long term outcomes of TAVI between males and females to try and identify specific tailored treatment options.

This data will be useful in providing important information regarding gender differences in patients who are treated with transcatheter aortic valve implantation. Data provided will include long term outcomes and predictors of outcome.

The study team will then identify and implement strategies to improve outcomes in patients being treated with transcatheter aortic valve implantation.

DETAILED DESCRIPTION:
Severe aortic stenosis (AS) is the commonest form of valvular abnormality in the developed world and accounts for more than 40% of patients with native valvular disease with an approximately equal prevalence in males and females.

Transcatheter aortic valve implantation (TAVI) is now widely practiced with treatment of over 300,000 patients worldwide. Many centres now regularly implant devices in patients for whom conventional aortic valve replacement (AVR) is deemed high or intermediate risk. Several studies have shown that females have an apparent better outcome with TAVI than males.

There are numerous possible reasons as to the apparent favourable benefit of TAVI in women including: having both lower rates of moderate / severe aortic regurgitation and peri-procedural mortality, lower rates of bleeding and renal failure, better patient prosthesis match and recovery of left ventricular function with more favourable left ventricular remodelling.

Rationale for proposal:

Newer devices have reduced the introducer French size and are hence associated with reduced rates of vascular and bleeding complications. This may translate to an even higher survival benefit in female versus male patients with severe aortic stenosis treated with transfemoral TAVI. In the current study we will aim to investigate gender temporal survival trends, and complications including stroke and heart attack in aortic stenosis patients treated with current versus older generation transcatheter valves. We have already been successful in obtaining the periprocedural data from NICOR and and mortality data will be linked from NHS digital.

Objectives

The current study will aim to:

1. Compare the mid-long term survival of females versus males in patients with AS treated with current versus older TAVI technologies. Study design In the current study, all patients undergoing transfemoral TAVI in the UK (between 2007 and 2017) will be included.

ELIGIBILITY:
All comers - retrospective registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All comers - national UK registry of all TAVI patients between 2007 - 2017
Sampling Method: Non-Probability Sample
Enrollment: 14086 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | 3 years
  Death
Cardiovascular Mortality | 3 years
  cardiac death

SECONDARY OUTCOMES:
Major adverse cardiovascular events | 3 years
  myocardial infarction, stroke, heart failure hospitalisations
Bleeding (according to BARC - life threatening, major, minor) | 3 years
  BARC classification

IPD SHARING:
Plan to Share IPD: No